CLINICAL TRIAL: NCT00003263
Title: Phase I Combined Modality Protocol for Malignant Mesothelioma: Cisplatin & rIFN-alpha-2b Followed by Surgical Resection (Debulking), and Post-Op Concurrent Chemoradiotherapy With Cisplatin, +/- rIFN-alpha-2b
Brief Title: Cisplatin, Interferon Alfa, Surgery, and Radiation Therapy in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Corey Langer, FCCC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066157; P30CA006927 (NIH); FCCC-96087; NCI-G98-1401
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Interferon-alpha; Cisplatin; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Biological: recombinant interferon alfa — vaccine
Drug: cisplatin
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Interferon alfa may interfere with the growth of cancer cells. Combining chemotherapy, radiation therapy, and interferon alfa may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of cisplatin plus interferon alfa followed by surgery and interferon alfa plus radiation therapy in treating patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of neoadjuvant interferon alfa 2b (IFN-A2b) administered with cisplatin in patients with malignant pleural mesothelioma. II. Determine the MTD of IFN-A2b administered with radiation therapy and cisplatin after surgery in these patients. III. Determine the response rate and toxicity of induction therapy with IFN-A2b and cisplatin in these patients. IV. Determine the toxicity of concurrent radiation therapy, cisplatin, and IFN-A2b after surgery in these patients. V. Determine the local control rate, freedom from progression, median survival, and long term survival of these patients after combined modality therapy.

OUTLINE: This is a dose escalation study. Patients receive induction therapy consisting of cisplatin IV weekly and interferon alfa 2b (IFN-A2b) subcutaneously three times a week for 6 weeks. Patients who experience at least 25% tumor shrinkage receive another 4 weeks of therapy. Patients then undergo debulking surgery to remove all gross tumor, if possible. If this resection is performed, then patients begin radiation therapy 2-6 weeks after surgery. Patients with unresectable tumors begin radiation therapy 2-4 weeks after the last course of induction chemotherapy. Patients undergo radiation therapy 5 days a week for 6 weeks. Concurrently, patients receive cisplatin IV weekly and IFN-A2b subcutaneously three times a week. Cohorts of 4 patients each receive escalated doses of IFN-A2b during induction chemotherapy. Once the maximum tolerated dose (MTD) of IFN-A2b is established, one dose level below this dose is used for the beginning doses of IFN-A2b during adjuvant chemotherapy. If no unacceptable toxic effects occur, then the dose of IFN-A2b is escalated to the induction MTD. Patients are followed at 3-6 weeks after completing radiochemotherapy, then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven ipsilateral malignant pleural mesothelioma
* No contralateral thoracic or intra-abdominal involvement
* No distant metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0 or 1
* Life expectancy: Not specified
* Hematopoietic:

  * Absolute neutrophil count greater than 2,000/mm3
  * Platelet count greater than 100,000/mm3
  * No symptomatic anemia requiring transfusion
* Hepatic:

  * Bilirubin less than 2.0 mg/dL
  * No autoimmune hepatitis
  * No history of decompensated liver disease; e.g. esophageal varices
  * Ascites
  * Albumin at least 2.5 mg/dL
  * Increasing prothrombin time of at least 2.0
* Renal: Creatinine no greater than 1.5 mg/dL
* Cardiovascular:

  * No symptomatic or debilitating cardiovascular disease,
  * No concurrent thrombophlebitic or embolic disorders
* Pulmonary:

  * No symptomatic or debilitating pulmonary disease,
  * Pretreatment diffusion capacity greater than 30% of predicted normal
  * Projected post-treatment FEV1 at least 1.0 L
* Other:

  * No prior malignancy within 3 years, except nonmelanomatous skin cancer
  * Carcinoma in situ of the cervix
  * Ductal carcinoma in situ of the breast
  * Not pregnant
  * Fertile patients must use effective contraception
  * No history of hypersensitivity to interferon or any component of the injection
  * No uncontrolled diabetes (blood sugars consistently at least 300 mg/dL)
  * No insulin dependent diabetes mellitus with history of ketoacidosis within 1 year
  * No psychosis
  * No uncontrolled thyroid abnormalities
  * No active infection requiring intravenous antibiotics

PRIOR CONCURRENT THERAPY:

* Biologic therapy: No prior biologic therapy
* Chemotherapy: No prior chemotherapy
* Endocrine therapy: Not specified
* Radiotherapy: No prior radiotherapy
* Surgery:

  * No prior debulking surgery
  * No prior chest tube drainage with sclerosis if tumor resectable
  * Prior thoracentesis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1996-08; Primary Completion 1999-12 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Office of S. Terry Kraus, Marrero, Louisiana
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Virginia Oncology Associates, Newport News, Virginia